CLINICAL TRIAL: NCT00933426
Title: A Modular Phase I-II Trial of Lenalidomide and Paclitaxel in Men With Castration-Resistant Prostate Cancer and Lymph-Node Dominant Metastases
Brief Title: Lenalidomide and Paclitaxel in Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated early due to slow accrual as Phase I dose escalation study.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0606; NCI-2010-01039 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
Keywords: Castration-Resistant Prostate Cancer; CRPC; Prostate; Lenalidomide; Revlimid; CC-5103; Paclitaxel; Taxol; Taxanes
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lenalidomide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide and Paclitaxel (Experimental): Phase I: Up to 5 differing doses of Lenalidomide tested plus fixed dose of Paclitaxel.
  Phase II: Lenalidomide at highest tolerated dose from Phase I plus Paclitaxel.
  Interventions: Drug: Lenalidomide; Drug: Paclitaxel

INTERVENTIONS:
Drug: Lenalidomide — Lead-In beginning dose of 5 mg capsules by mouth once a day for 21 days in a row, followed by 7 days of rest (Days 22-28) for a 28 day cycle.
  Other Names: Revlimid; CC-5013
Drug: Paclitaxel — 50 mg/m^2 given by vein over 1 hour on Days 1, 8, and 15 of each 28 day cycle.
  Other Names: Taxol

SUMMARY:
The goal of the Phase I part of this clinical research study is to find the highest tolerable dose of Revlimid® (lenalidomide) that can be given in combination with paclitaxel to patients with prostate cancer who have failed treatment with taxanes.

The goal of the Phase II part of this clinical research study is to learn if lenalidomide and paclitaxel can help to control prostate cancer.

The safety of this combination treatment will be studied in both phases of the study.

UPDATE:

Study was terminated early due to slow accrual as a Phase I dose escalation study, without progression to Phase II study portion.

DETAILED DESCRIPTION:
Study Drugs:

Lenalidomide is a drug that changes the immune system and it may also interfere with the development of tiny blood vessels that help support tumor growth. Taking lenalidomide could prevent the growth of cancer cells.

Paclitaxel is designed to disrupt the growth of cancer cells, which may cause cancer cells to die.

Phases I and II:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you joined the study. Up to 10 groups of 3 participants will be enrolled in the Phase I portion of the study, and 1 group of up to 42 participants will be enrolled in Phase II.

If you are enrolled in the Phase I portion, the doses of lenalidomide you receive will depend on when you joined this study. The dose of paclitaxel will be the same for all patients. Up to 5 dose levels of lenalidomide will be tested in the Phase I portion. The first group of Phase I participants will receive the lower doses of lenalidomide. Each new group enrolled will receive the higher doses, if no intolerable side effects were seen. Groups will continue being enrolled (up to 10) until the highest tolerable dose of lenalidomide (in combination with paclitaxel) is found.

If you are enrolled in the Phase II portion, you will receive lenalidomide at the highest dose that was tolerated in the Phase I portion in combination with paclitaxel.

Study Drug Administration:

Once you are assigned a dose, you will take lenalidomide capsules by mouth once a day for 21 days in a row, followed by 7 days of rest (Days 22-28). This will be called the "lead-in" period."

You will the begin taking lenalidomide and paclitaxel on 28 day study cycles. You will take lenalidomide by mouth every day on Days 1-21 of each cycle. Paclitaxel will be given by vein over 1 hour on Days 1, 8, and 15 of each cycle. On Days 22-28 of each cycle, you will take no study drugs. The Day 1 dose of Lenalidomide in each combination cycle may occur within +/- 5 days of the Day 1 paclitaxel dose.

You should swallow lenalidomide capsules whole with water at the same time each day. Do not break, chew, or open the capsules.

If you miss a dose of lenalidomide, take it as soon as you remember on the same day.

If you miss taking your dose for the entire day, take your regular dose the next scheduled day (do NOT take double your regular dose to make up for the missed dose).

If you take more than the prescribed dose of lenalidomide you should seek emergency medical care, if needed, and contact study staff right away.

Females of childbearing potential that might be caring for you should not touch the lenalidomide capsules or bottles unless they are wearing gloves.

In order to participate in this study you must also register into and follow the requirements of the RevAssist® program of Celgene Corporation. This program provides education and counseling on the risks of fetal exposure, blood clots, and reduced blood counts. You will be required to receive counseling every 28 days during treatment with lenalidomide, follow the birth control requirements of the program that are appropriate for you, and take telephone surveys about your compliance with the program.

Study Visits:

On Day 1 of each cycle (before you receive paclitaxel), the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight.
* Your performance status will be recorded.
* You will be asked about any drugs or treatments you may be receiving.
* Blood (about 2-3 teaspoons) will be drawn for routine tests and tests of your prostatic specific antigen (PSA) and testosterone levels.
* You will be asked about any side effects you may have experienced since your last visit.

On Days 8 and 15 of each cycle (before you receive paclitaxel), the following tests and procedures will be performed:

* Your weight will be measured.
* Blood (about 2 teaspoons) will be drawn for routine tests.

On Day 1 of Cycle 3 and every 2 cycles thereafter, you will have the following tests and procedures performed:

* You will have a chest x-ray and a CT scan of your abdomen and pelvis to check the status of the disease.
* Blood (about 2 teaspoons) will be drawn to test your testosterone level and your liver function.
* You will have a bone scan to check the status of the disease.
* You will have an ECG.

If you are being treated with paclitaxel at your local oncologist's office, you are only required to return to M. D. Anderson on Days 1 and 15 of Cycle 1 and on Day 1 of each cycle after that. All other study visits may be done at your local oncologist's office.

Length of Study:

You will continue on this study as long as you are benefiting. You will be removed from the study if you experience intolerable side effects, if the disease gets worse, or if the study doctor thinks it is in your best interest.

End-of-Study Visit:

Once you are off study, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 3-4 teaspoons) will be drawn for routine tests and tests of your PSA and testosterone levels.
* You will be asked about any side effects you may have experienced since your last visit.
* Your performance status will be recorded.

This is an investigational study. Lenalidomide is approved by the Food and Drug Administration (FDA) and commercially available for the treatment of specific types of myelodysplastic syndrome (MDS) and in combination with dexamethasone for patients with multiple myeloma (MM) who have received at least 1 prior therapy. Paclitaxel is FDA-approved and commercially available for the treatment of bladder cancer, lung cancer, breast cancer, and pancreatic cancer. The use of these drugs in combination is investigational.

Up to 72 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic adenocarcinoma of the prostate
2. Patients in Phase II must have radiographic evidence of multiple (>/= 2) or bulky (>/= 5cm diameter) lymph node metastases with < 2 bone (on radionuclide bone scan) discrete sites of involvement.
3. Patient must have had front-line chemotherapy for castrate-resistant metastatic disease. Any number of prior chemotherapy regimens is permitted, except within the last 3 weeks. No prior thalidomide or lenalidomide therapy is permitted.
4. Patients must have evidence of progression of disease based on any one of the following criteria: a) PSA- progression is defined as 2 consecutive increments in PSA (with an absolute change of at least 1ng/mL) over 4 weeks. b) An increase by 25% of the product of bi-dimensional disease or 30% in maximum diameter or appearance of an unequivocally new lesion qualifies as progression. c) Worsening symptoms clearly attributable to disease progression qualifies as progression e.g. worsening malignant bony pain.
5. Patients on antiandrogens should be discontinued from flutamide, nilutamide or cyproterone acetate for at least 4 weeks and bicalutamide for 6 weeks. If progression is documented during or after this time interval, patients are eligible. Patients who have not had response to deferred (secondary) therapy with antiandrogens do not have to satisfy this waiting period prior to enrollment.
6. Patients must have a performance status of </= 2 (ECOG).
7. Patients will not receive any concurrent biological, immunological, second-line hormonal therapy or chemotherapy. Patients receiving replacement or therapeutic doses of corticosteroid for non-malignant disease while disease progression was established may continue on such therapy.
8. Patients must have recovered from prior chemotherapy, biological or immunological therapy or radiation delivered within the last 28 days. Radioisotope therapy with strontium delivered within the last 90 days or samarium within the last 60 days is not permitted.
9. Patients must have a castrate serum testosterone level (</= 50ng/ml) documented in the last six weeks. For patients who are medically castrated, luteinizing hormone releasing hormone analog must continue to maintain testicular suppression.
10. Patients must have adequate bone marrow function defined as an absolute peripheral granulocyte count of >/= 1,500/mm^3 and platelet count of >/= 75,000/mm^3.
11. Patients must have adequate hepatic function defined with a bilirubin of </= 2 X upper limits of normal and AST/ALT </= 2.5 X the upper limits of normal.
12. Patients must have adequate renal function defined as creatinine clearance >/= 40 cc/min (measured or calculated by Cockcroft and Gault formula).
13. Must be fully recovered from any previous surgery, in terms of wound healing.
14. Patients must sign an informed consent indicating that they are aware of the investigational nature of this study, in keeping with the policies of the institution.
15. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
16. Men must agree to use a latex condom during sexual contact with a female of childbearing potential (FCBP) even if they have had a successful vasectomy. A FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
17. Patient must be able to take low molecular weight heparin (preferred) OR low-dose enteric aspirin and warfarin for thromboembolic prophylaxis.

Exclusion Criteria:

1. Patients with severe or uncontrolled infection defined as symptomatic and/or requiring intravenous antibiotics.
2. Patients with small cell or sarcomatoid variant of prostate cancer.
3. Patients with symptomatic congestive heart failure (CHF), pulmonary embolus, vascular thrombosis, transient ischemic attack, cerebrovascular accident, unstable angina or MI in the last 3 months or evidence of active myocardial ischemia by symptoms or electrocardiogram (ECG).
4. Known severe hypersensitivity to taxanes.
5. Patients with central nervous system (CNS) metastasis or cord compression are excluded except those patients that have had complete excision or radiotherapy and remain asymptomatic for at least 2 months.
6. Oxygen-dependent lung disease or >/= grade 2 peripheral neuropathy.
7. Known intolerance of corticosteroid therapy that would preclude its use as premedication for paclitaxel.
8. Uncontrolled severe hypertension or uncontrolled diabetes mellitus.
9. Active second malignancies. Non-threatening second malignancies such as superficial low-grade transitional cell carcinoma of the bladder or Rai Stage 0 chronic lymphocytic leukemia or stable small renal cell carcinomas may be exempt from such stipulation at the discretion of the Principal Investigator.
10. Overt psychosis or mental disability or otherwise incompetent to give informed consent. Patients who are unwilling or unable to comply with the RevAssist® program or with a history of non-compliance with medical regimens or who are considered potentially unreliable.
11. Patients with known HIV or active hepatitis A, B, or C infection.
12. Patients receiving any concurrent biological, immunological, second-line hormonal therapy or chemotherapy. Patients receiving replacement or therapeutic doses of corticosteroid for non-malignant disease while disease progression was established may continue on such therapy.
13. Patients who have not recovered from prior chemotherapy, biological or immunological therapy or radiation delivered within the last 28 days. Radioisotope therapy with strontium delivered within the last 90 days or samarium within the last 60 days is not permitted.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of Lenalidomide in Combination with Low-Dose Weekly Paclitaxel | After 2, 28 day cycles
  MTD defined as dose with posterior mean Pr{toxicity} closest to .33 at the end of the trial, provided that it is not terminated early. The CRM will be implemented using fixed toxicity probabilities (p1, p2, p3, p4, p5) = (.05, .20, .33, .45, .60) under the model Pr{toxicity | dose level j} = {pj}exp(a) , where a follows a normal prior with mean 0 and variance 2. Dose limiting toxicity (DLT) defined as any of the following treatment-related events occurring within two cycles of therapy (i) uncontrolled or intolerable grade 2 non-hematologic toxicity > 7 days, (ii) grade 3or 4 nausea/vomiting/diarrhea > 48 hours, (iii) > grade 3 fatigue > 7 days and any other grade 3or 4 non-hematologic toxicity; (iv) grade 4 hematologic toxicity (v) neutropenic fever defined as absolute neutrophil count (ANC) < 1000 and temperature >/ 101 degrees F; (vi) any other regimen-related adverse event that precludes delivery of the first two cycles of therapy.

SECONDARY OUTCOMES:
Progression-Free (PFS) Time in Patients with a Lymph Node Dominant Clinical Phenotype | After 2, 28 day cycles
  The unadjusted PFS time distribution estimated using method of Kaplan and Meier. A Cox model or other appropriate time-to-event regression model, chosen based on preliminary goodness-of-fit analyses, used to assess the ability of either baseline or change during lead-in in biomarker status, as well as conventional covariates including performance status, hemoglobin and LDH, to predict PFS.
  13.0

CONTACTS AND LOCATIONS:
Overall Officials: Lance Pagliaro, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org